CLINICAL TRIAL: NCT05303337
Title: Evolution of HIV Reservoir, Inflammation and Microbiota Footprint of PLWH Switching to Long-acting Injectable Treatment Compared to Patients on Oral Dual or Triple Anti-integrase-based Therapy: a Prospective Longitudinal Comparative Study
Brief Title: Evolution of HIV Reservoir, Inflammation and Microbiota Footprint of PLWH Switching to Long-acting Injectable Treatment Compared to Patients on Oral Dual or Triple Anti-integrase-based Therapy
Acronym: LAMIVIH
Status: Recruiting | Type: Observational
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 21-40
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients switching towards a long-aging injectable treatment
  Interventions: Other: Stool sampling; Other: Blood plasma collection
- Patients maintaining oral ART 2-drug regimens
  Interventions: Other: Stool sampling; Other: Blood plasma collection
- Patients maintaining oral ART 3 drug regimens
  Interventions: Other: Stool sampling; Other: Blood plasma collection

INTERVENTIONS:
Other: Stool sampling — Stool samples will be collected from participants at baseline and W52
Other: Blood plasma collection — Blood plasma collection to assess persistent inflammation, immune activation and HIV reservoir at baseline,W24,W52

SUMMARY:
In the last 40 years of HIV history, we have managed to attain most of our therapeutic objectives, namely virological suppression of most patients and sufficient immune reconstitution. Still, immune activation and inflammation persist and even if they decrease on ART (AntiRetroviral Treatment), they do not disappear and may be associated to multiple non-AIDS related comorbidities.

In this population structural and functional modifications of GALT (Gut Associated Lymphoïd Tissue) are observed early after HIV infection and persist despite virological suppression on ART. Moreover, imbalance of the gut microbiota which is called dysbiosis may participate in persistent activation and therefore enhancement of residual HIV viral replication.

GALT modifications are associated with microbial translocation that is also correlated with immune activation and dysbiosis.

Up to now, there is no evidence of a differential impact on inflammation, immune activation or cellular reservoirs of different ART regimens. Long-Acting (LA) regimens could theoretically display better inflammatory profile, since they have a better tissue distribution and could act more efficiently on HIV reservoirs. On the other hand, LA's direct administration shunting the gut passage could also contribute to less gut dysbiosis.

The objective of our study is to assess impact on plasma biomarkers, cell-surface biomarkers, intestinal microbiota and cellular reservoirs of a switch from an oral dual or triple anti-integrase-based therapy ART regimen including an anti-integrase compared to a Long-Acting (LA) injectable treatment.

ELIGIBILITY:
Inclusion Criteria:

* PLWH at a the stable phase of their disease (absence of disease outbreak and absence of treatment modification in the 3 months preceding inclusion),
* Subject with ongoing HIV follow-up on an outpatient basis (outpatient or day hospital consultation) in the participating center, and having virological suppression at the threshold of 50 copies / mL for at least 1 year (blips < 200 copies / mL tolerated during this period)
* CD4 + T cell nadir> 200 / mm3
* Having given free and informed written consent
* Being affiliated with or benefiting from a social security scheme.

Exclusion Criteria:

* Persons treated with antibiotics, probiotics, prebiotics or any other treatment that may disrupt the gut microbiota within two month before stool sampling.
* Subject only coming for full impatient follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People Living with HIV (PLWH)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Variation of the HIV cellular reservoirs at W52 of two switch comparatively to baseline among the 3 groups of PLWH | 12 months

SECONDARY OUTCOMES:
Variation of the Shannon index between 0 and 1 year in the different groups of PLWH compared to baseline | 12 months
Variation of the immune profile in participants with an LA-based regimen compared to participants with an oral therapy at W24 and W52 | 12 months
Correlation between the immune profile and the Shannon index at W52 among the different groups of PLWH | 12 months
Correlation between the immune profile and the HIV-reservoirs at W52 among the different groups of PLWH | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Marseille, Marseille, France